CLINICAL TRIAL: NCT05181202
Title: Biomarkers Study of Liposomal Doxorubicin Injection Induced Hypersensitivity Reaction in Breast Cancer Patients
Brief Title: Biomarkers of Liposomal Doxorubicin Induced Hypersensitivity Reaction in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: YDPLD191016-I1-SYSU-001
Record Dates: First submitted 2021-12-21; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Liposomal Doxorubicin Induced Hypersensitivity Reaction in Breast Cancer Patients
Keywords: liposomal doxorubicin; hypersensitivity reaction; breast cancer
MeSH Terms: conditions — Hypersensitivity; Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hypersensitivity reaction group: The patients get hypersensitivity after Pegylated liposomal doxorubicin injection.
  Interventions: Other: Blood sampling
- None hypersensitivity reaction group: The patients do not get hypersensitivity after Pegylated liposomal doxorubicin injection.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Collect blood before drug injection. we do not intervene the clinical administration or drug choice or other clinical treatment.

SUMMARY:
Pegylated liposomal doxorubicin (PLD) was an anthracycline nanomedicine to be approved for advanced breast cancer and other solid tumor therapy and showed a good disease control rate (57%). PLD could induce hypersensitivity reaction (HSR). There are about 9-25% patients got infusion reaction or HSR. Severe HSR could lead to allergic shock even presyncope or threat to life. To our knowledge, there were no sensitivity biomarker to predict the PLD induced HSR. And the mechanism of PLD induced HSR is unknown yet. Therefore, to analyze and discuss the biomarkers and mechanism of PLD induced HSR in advanced breast cancer, we design this prospective, observational, biomarker study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old; Breast cancer confirmed with histological or molecular diagnosis; Advanced breast cancer diagnosis according to American Joint Committee on cancer eighth edition cancer staging manual; Treatment with liposomal doxorubicin; No pregnancy plan and voluntary use of effective contraceptive measures during treatment

Exclusion Criteria:

* Subjects who discontinued treatment due to previous severe adverse reactions to liposomal doxorubicin or doxorubicin; poor compliance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced breast cancer patients who recieve liposomal doxorubicin treatment.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The predictive biomarkers of PLD induced hypersensitivity | 2022.06-2023.12
  Detect and analyze the association between hypersensitivity and metabonomics, anti-PEG antibody, IgE et. al

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
If we found a significant, sensitive biomarker of liposomal doxorubicin induced hypersensitivity, we will share the protocol and results with other scientists or clinical researchers.

REFERENCES:
- [Background] Alberts DS, Garcia DJ. Safety aspects of pegylated liposomal doxorubicin in patients with cancer. Drugs. 1997;54 Suppl 4:30-5. doi: 10.2165/00003495-199700544-00007. PMID 9361959
- [Background] Castells MC, Tennant NM, Sloane DE, Hsu FI, Barrett NA, Hong DI, Laidlaw TM, Legere HJ, Nallamshetty SN, Palis RI, Rao JJ, Berlin ST, Campos SM, Matulonis UA. Hypersensitivity reactions to chemotherapy: outcomes and safety of rapid desensitization in 413 cases. J Allergy Clin Immunol. 2008 Sep;122(3):574-80. doi: 10.1016/j.jaci.2008.02.044. Epub 2008 May 27. PMID 18502492
- [Background] Chen E, Chen BM, Su YC, Chang YC, Cheng TL, Barenholz Y, Roffler SR. Premature Drug Release from Polyethylene Glycol (PEG)-Coated Liposomal Doxorubicin via Formation of the Membrane Attack Complex. ACS Nano. 2020 Jul 28;14(7):7808-7822. doi: 10.1021/acsnano.9b07218. Epub 2020 Mar 6. PMID 32142248
- [Background] Gabizon A, Szebeni J. Complement Activation: A Potential Threat on the Safety of Poly(ethylene glycol)-Coated Nanomedicines. ACS Nano. 2020 Jul 28;14(7):7682-7688. doi: 10.1021/acsnano.0c03648. Epub 2020 Jul 9. PMID 32643376
- [Background] Verhoef JJ, Carpenter JF, Anchordoquy TJ, Schellekens H. Potential induction of anti-PEG antibodies and complement activation toward PEGylated therapeutics. Drug Discov Today. 2014 Dec;19(12):1945-52. doi: 10.1016/j.drudis.2014.08.015. Epub 2014 Sep 7. PMID 25205349
- See also: breast cancer epidemiology — https://gco.iarc.fr/today/data/factsheets/cancers/20-Breast-fact-sheet.pdf